CLINICAL TRIAL: NCT03168672
Title: GLOBAL ICON Stemless Shoulder System Post Market Clinical Follow Up Study
Acronym: Global ICON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of concerns about subject attrition between the 5- and 10-year visits. A nested PMCF study at 10 years was proposed to the regulatory body and it was agreed this was an acceptable approach
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 1401
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Post Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Global ICON (Other): The study device is the GLOBAL ICON stemless humeral component, consisting of the Anchor Plate and Humeral Head.
  Interventions: Device: Global ICON

INTERVENTIONS:
Device: Global ICON — The study device is the GLOBAL ICON stemless humeral component, consisting of the Anchor Plate and Humeral Head.

SUMMARY:
This is a Post Market Clinical Follow Up (PMCF) study to monitor the safety and performance of the GLOBAL ICON stemless humeral component. The data gathered will be used to support post market surveillance of the device, and may potentially be used for additional market access purposes.

DETAILED DESCRIPTION:
This study will be multi-centre and non-comparative. Subjects will be recruited and followed up at similar intervals to reflect the standard clinical practice and intended population for wider use of the device.

157 non-randomised subjects will be recruited from approximately 15 sites. A maximum of 30 subjects may be recruited from one site. More than one implanting surgeon may recruit subjects at each site as a designated sub-Investigator.

The primary objective of this PMCF study is to confirm device survivorship of the GLOBAL ICON stemless humeral component at 24 months post-operative.

The secondary objectives include the evaluation of clinical performance, radiographic performance and safety outcomes at 3, 12, 24, 60 and 120 months post-operatively.

Tertiary endpoints in the study will include a mean change from baseline for the Adjusted Constant-Murley Score, the Oxford Shoulder Score, the EQ-5D-5L dimension score and EQ-VAS scores. Radiographic evidence of aseptic loosening and periprosthetic fracture survivorship of the GLOBAL ICON stemless humeral component will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Severely painful and/or severely disabled Non-Inflammatory Degenerative Joint Disease (NIDJD) resulting from osteoarthritis (OA) or post traumatic arthritis Patient is willing and able to complete the required post-operative schedule Patient has provided written Informed Consent to participate

Exclusion Criteria:

Subjects under the age of 21 or over the age of 80 on the day of consent Subjects who have not reached skeletal maturity, regardless of age Inadequate bone stock in the proximal humerus or glenoid fossa for supporting the GLOBAL ICON stemless humeral components Bone that is too soft or porous to support the implant or that is too hard or brittle to allow for proper bone preparation and fixation, i.e osteoporosis or sclerotic bone, where there could be considerable migration of the prosthesis and/or a chance of fracture of the humerus or glenoid Fractures of the proximal humerus that could compromise the fixation of the GLOBAL ICON stemless humeral components Subjects who have undergone previous treatment on the study shoulder that may compromise fixation of the GLOBAL ICON stemless humeral components Revision of a failed hemi, total or reverse shoulder arthroplasty Active local or systemic infection Absent, irreparable or nonfunctional rotator cuff or other essential muscles Subject is receiving, or is scheduled to receive, treatment that the Investigator considers could affect bone quality, such as chemotherapy or high dose corticosteroids Subjects who, at the point of enrolment, already have a GLOBAL ICON shoulder replacement or are scheduled to receive, a contralateral shoulder replacement device Subjects who are known to be pregnant or breastfeeding Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes Subjects with a known medical condition that the Investigator believes would impact the study outcomes (including, but not limited to osteomyelitis, Paget's disease, neuropathies such as Charcot's disease, metastatic or neoplastic disorders) Known polyethylene and/or metal sensitivity or allergy

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Kingston General Hospital, Kingston, Canada
- Germany (3):
  - Vulpius Klinik, Bad Rappenau
  - Orthopädische Klinik der Medizinischen Hochschule Hannover im Diakovere Annastift, Hanover
  - Sportklinik Ravensburg, Ravensburg
- Netherlands (3):
  - Treant Hospital, Emmen
  - Groene Hart Ziekenhuis, Gouda
  - Tergooi Hospital, Hilversum
- United Kingdom (5):
  - Woodend Hospital, Aberdeen
  - The Royal Bournemouth Hospital, Bournemouth
  - North Bristol NHS Trust, Bristol
  - James Cook University Hospital, Middlesbrough
  - City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for recruitment into the study from the general diagnosis population defined as total shoulder arthroplasty (TSA). The investigation was conducted at 12 centers.
Units Other Than Participants: Shoulders
Groups:
- GLOBAL ICON Stemless Shoulder System: Study participants who received a GLOBAL ICON Stemless shoulder system.
Period: Overall Study
Arm/Group | GLOBAL ICON Stemless Shoulder System
Started (172 shoulders from 171 participants were enrolled in the study. 156 participants received 157 implants (1 participant had staged bilateral shoulder surgery)) | 171; 172 Shoulders
Safety Population | 156; 157 Shoulders
Treated With GLOBAL ICON | 156; 157 Shoulders
Completed | 0; 0 Shoulders
Not Completed | 171; 172 Shoulders
Not completed — Withdrawal by Subject | 13
Not completed — Death | 3
Not completed — Investigator's Decision | 137
Not completed — Adverse Event | 1
Not completed — Other | 2
Not completed — Started but not treated with GLOBAL ICON | 15

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so.
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Study participant age (mean) | 66.0 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender of study participants: Female | 80
  Gender of study participants: Male | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Composite Clinical Success
Description: Percentage of participants with overall composite clinical success at 24 months was reported. Composite success was achieved if each of the following criteria was met: (1) Radiographs indicated that there was no continuous radiolucent line (RLL) around the GLOBAL ICON stemless humeral component, with continuous RLL defined as a radiolucent line greater than (>) 1millimeter (mm) in all five zones of either anterior-posterior (AP) or Axillary views (2) The adjusted Constant-Murley score was greater than 85, with the adjustment based on the method of Constant (3) No GLOBAL ICON humeral component was removed for any reason (4) There was no device-related serious adverse events.
Time Frame: At 24 months
Population: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 140
Percentage of participants | 82.86

2. Primary Outcome: Adjusted Constant-Murley Shoulder Assessment Score
Description: Constant-Murley Score on operative shoulder adjusted for gender and age. Please note that scores are adjusted to reflect gender and age of participants. The Constant-Murley score is divided into four subscales, including pain (15 points maximum), activities of daily living (20 points maximum), ROM (40 points maximum), and strength (25 points maximum). The higher the score, the higher the quality of function (minimum 0, maximum 100) Adjustment may lead to scores above 100 depending on age of group analyzed. The range for the Adjusted Constant-Murley score in a male participant is 0-178.6; the range for the Adjusted Constant-Murley score in a female participant is 0-192.3. Please note the calculations of the maximum Adjusted score assume a perfect score (100) in 100 year old male and female participants.
Time Frame: 24 Months
Population: Study participants who received a GLOBAL ICON Shoulder system.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Implants
Groups:
- GLOBAL ICON Stemless Shoulder Group: Participants who received a GLOBAL ICON Stemless Shoulder. Constant-Murley Score on operative shoulder adjusted for gender and age. Please note that scores are adjusted to reflect gender and age of participants. The Constant-Murley score is divided into four subscales, including pain (15 points maximum), activities of daily living (20 points maximum), ROM (40 points maximum), and strength (25 points maximum). The higher the score, the higher the quality of function (minimum 0, maximum 100) Adjustment may lead to scores above 100 depending on age of group analyzed.
Arm/Group | GLOBAL ICON Stemless Shoulder Group
Number analyzed (Participants) | 138
Number analyzed (Implants) | 138
Units on a scale | 103.7 (21.8)

3. Primary Outcome: Continuous Radiolucent Line
Description: X-rays are reviewed by an independent radiographic reviewer to determine if a 1 mm wide or greater, continuous radiolucent line around the entire bony border of the GLOBAL ICON Stemless Shoulder implant exists. Such a line may indicate the implant is loosening.
Time Frame: 24 months
Population: All participants who received a GLOBAL ICON Stemless Shoulder were evaluated radiographically at 24 months for the presence of a continuous radiolucent line around the implant that was greater than 1mm wide.
Measure: Count of Participants; unit: Participants
Groups:
- GLOBAL ICON Stemless Shoulder Group: Study participants who received a GLOBAL ICON Stemless Shoulder Implant.
Arm/Group | GLOBAL ICON Stemless Shoulder Group
Number analyzed (Participants) | 142
Participants | 0

4. Primary Outcome: Kaplan Meier Survivorship
Description: Kaplan Meier Survival Estimate is based upon the number of GLOBAL ICON implants remaining in the study and the number of GLOBAL ICON implants that have been revised (surgically removed from participants).
Time Frame: 24 months
Population: Study participants who received a GLOBAL ICON Shoulder System.
Measure: Number (95% Confidence Interval); unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | GLOBAL ICON Stemless Shoulder Group
Number analyzed (Participants) | 120
Number analyzed (Implants) | 120
Percentage of implants | 98.7 [95.0 to 99.7]

5. Primary Outcome: Device-related Serious Adverse Events
Description: Adverse events are any untoward health issues that occur when compared to a participant's normal health baseline. Serious adverse events include health events that have led to death or a serious deterioration in health that resulted in life threatening illness/injury, permanent impairment of a body structure, required hospitalization or required medical intervention to prevent life threatening illness/injury or permanent impairment to a body structure or function.
Time Frame: 24 months
Population: Study participants who received a GLOBAL ICON shoulder system
Measure: Count of Participants; unit: Participants
Arm/Group | GLOBAL ICON Stemless Shoulder Group
Number analyzed (Participants) | 156
Participants | 1

6. Secondary Outcome: Mean Adjusted Constant-Murley Score at Baseline, 3, 12, 24, and 60 Months Post-operative
Description: Constant-Murley Score was adjusted to reflect gender and age of participants. The Constant-Murley score was divided into four subscales, including pain (15 points maximum), activities of daily living (20 points maximum), ROM (40 points maximum), and strength (25 points maximum). The higher the score, the higher the quality of function (minimum 0, maximum 100). Adjustment may lead to scores above 100 depending on age of group analyzed. The range for the Adjusted Constant-Murley score in a male participant was 0-178.6; the range for the Adjusted Constant-Murley score in a female participant was 0-192.3. The calculations of the maximum Adjusted score assume a perfect score (100) in 100 year old male and female participants.
Time Frame: At Baseline (Day 0), 3, 12, 24, and 60 months
Population: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so. Here, n (number analyzed) signifies number participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Unit on a scale
  Baseline | 42.2 (22.5)
  3 Months: number analyzed (Participants) | 152
  3 Months | 70.0 (23.1)
  12 Months: number analyzed (Participants) | 130
  12 Months | 95.5 (22.8)
  24 Months: number analyzed (Participants) | 138
  24 Months | 103.7 (21.7)
  60 Months: number analyzed (Participants) | 123
  60 Months | 106.2 (21.7)

7. Secondary Outcome: Mean Oxford Shoulder Score at Baseline, 3, 12, 24, and 60 Months Post-operative
Description: The Oxford Shoulder Score (OSS) was a patient-based questionnaire used to assess shoulder pain after surgery. It consisted of 12 questionnaire items with 5 ordinal response options for each question. Each response was scored from 0 to 4 points (4 = best/least problems and 0=worst/unbearable pain). All item scores across 12 questions were summed to produce a scale of 0-48 (where a higher score reflected best/least problems).
Time Frame: At Baseline (Day 0), 3, 12, 24, and 60 months
Population: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so. Here, n (number of participants analyzed) signifies number participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Unit on a Scale
  Baseline | 20.6 (8.2)
  3 Months: number analyzed (Participants) | 153
  3 Months | 35.1 (9.8)
  12 Months: number analyzed (Participants) | 129
  12 Months | 41.9 (7.7)
  24 Months: number analyzed (Participants) | 137
  24 Months | 43.1 (7.4)
  60 Months: number analyzed (Participants) | 123
  60 Months | 43.5 (7.6)

8. Secondary Outcome: Mean EuroQol-5 Dimension 5-Level (EQ-5D-5L) Scores by Dimensions at Baseline, 3, 12, 24, and 60 Months Post-operative
Description: Mean EQ-5D-5L scores by dimensions at baseline, 3, 12, 24, and 60 months were reported. EQ-5D-5L consisted of the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ-VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5-item index score was transformed into a utility score between 0 (worst health state) and 1 (best health state). Higher score indicated good health. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicated improvement.
Time Frame: At Baseline (Day 0), 3, 12, 24, and 60 months
Population: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so. Here, n (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Unit on a Scale
  Mobility: Baseline | 1.8 (1.04)
  Mobility: 3 Months: number analyzed (Participants) | 152
  Mobility: 3 Months | 1.5 (0.90)
  Mobility: 12 Months: number analyzed (Participants) | 129
  Mobility: 12 Months | 1.6 (0.93)
  Mobility: 24 Months: number analyzed (Participants) | 137
  Mobility: 24 Months | 1.7 (0.99)
  Mobility: 60 Months: number analyzed (Participants) | 123
  Mobility: 60 Months | 1.7 (0.97)
  Self-Care: Baseline | 2.4 (1.02)
  Self-Care: 3 Months: number analyzed (Participants) | 153
  Self-Care: 3 Months | 1.6 (0.87)
  Self-Care: 12 Months: number analyzed (Participants) | 129
  Self-Care: 12 Months | 1.3 (0.61)
  Self-Care: 24 Months: number analyzed (Participants) | 137
  Self-Care: 24 Months | 1.3 (0.61)
  Self-Care: 60 Months: number analyzed (Participants) | 123
  Self-Care: 60 Months | 1.3 (0.67)
  Usual Activities: Baseline | 3.0 (1.00)
  Usual Activities: 3 Months: number analyzed (Participants) | 153
  Usual Activities: 3 Months | 2.0 (0.97)
  Usual Activities: 12 Months: number analyzed (Participants) | 129
  Usual Activities: 12 Months | 1.6 (0.85)
  Usual Activities: 24 Months: number analyzed (Participants) | 137
  Usual Activities: 24 Months | 1.5 (0.87)
  Usual Activities: 60 Months: number analyzed (Participants) | 123
  Usual Activities: 60 Months | 1.6 (0.83)
  Pain/Discomfort: Baseline | 3.5 (0.82)
  Pain/Discomfort: 3 Months: number analyzed (Participants) | 152
  Pain/Discomfort: 3 Months | 2.2 (0.80)
  Pain/Discomfort: 12 Months: number analyzed (Participants) | 129
  Pain/Discomfort: 12 Months | 2.0 (0.94)
  Pain/Discomfort: 24 Months: number analyzed (Participants) | 137
  Pain/Discomfort: 24 Months | 1.9 (0.97)
  Pain/Discomfort: 60 Months: number analyzed (Participants) | 123
  Pain/Discomfort: 60 Months | 2.1 (1.01)
  Anxiety/Depression: Baseline | 1.7 (0.98)
  Anxiety/Depression: 3 Months: number analyzed (Participants) | 152
  Anxiety/Depression: 3 Months | 1.4 (0.76)
  Anxiety/Depression: 12 Months: number analyzed (Participants) | 129
  Anxiety/Depression: 12 Months | 1.4 (0.75)
  Anxiety/Depression: 24 Months: number analyzed (Participants) | 137
  Anxiety/Depression: 24 Months | 1.4 (0.78)
  Anxiety/Depression: 60 Months: number analyzed (Participants) | 123
  Anxiety/Depression: 60 Months | 1.3 (0.66)

9. Secondary Outcome: Mean Visual Analog Scale (EQ-VAS) Score at Baseline, 3, 12, 24, and 60 Months Post-operative
Description: EQ-5D-5L consisted of the EQ-5D-5L descriptive system and the EQ-VAS. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicated improvement.
Time Frame: At Baseline (Day 0), 3, 12, 24, and 60 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Unit on a scale
  Baseline | 64.7 (21.9)
  3 Months: number analyzed (Participants) | 153
  3 Months | 75.6 (15.8)
  12 Months: number analyzed (Participants) | 129
  12 Months | 78.1 (17.6)
  24 Months: number analyzed (Participants) | 138
  24 Months | 79.3 (16.3)
  60 Months: number analyzed (Participants) | 123
  60 Months | 78.0 (17.6)

10. Secondary Outcome: Number of Participants With Radiographic Evidence of Aseptic Loosening of the Global Icon Stemless Humeral Component Immediate Post-operative and 3, 12, 24, and 60 Months Post-operative
Description: Number of participants with radiographic evidence of aseptic loosening of the global icon stemless humeral component immediate post-operative and 3, 12, 24 and 60 months post-operative were reported. Aseptic Loosening was evaluated using all available imaging. Progressing radiolucencies and/or stress shielding indicated aseptic loosening.
Time Frame: Immediate post operative (0-10 Days), at 3, 12, 24, and 60 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GLOBAL ICON Stemless Shoulder System
Number analyzed (Participants) | 156
Participants
  Immediate Post Operative | 0
  3 Months: number analyzed (Participants) | 153
  3 Months | 0
  12 Months: number analyzed (Participants) | 131
  12 Months | 0
  24 Months: number analyzed (Participants) | 143
  24 Months | 0
  60 Months: number analyzed (Participants) | 122
  60 Months | 0

ADVERSE EVENTS:
Time Frame: Day 0 (Day of surgery) up to 60 months
Description: All-Cause Mortality: Analysis population included all enrolled participants. For SAEs and Non-SAEs: Safety population included all participants who were enrolled and were either implanted with the GLOBAL ICON stemless humeral component or an attempt was made to do so.
Arm/Group | GLOBAL ICON Stemless Shoulder System
All-Cause Mortality (participants affected / at risk) | 3/171
Serious Adverse Events (participants affected / at risk) | 75/156
Other Adverse Events (participants affected / at risk) | 100/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLOBAL ICON Stemless Shoulder System (N=156)
Acute myocardial infarction (Cardiac disorders) | 1 (6)
Angina pectoris (Cardiac disorders) | 1 (6)
Atrial fibrillation (Cardiac disorders) | 4 (6)
Glaucoma (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 1 (6)
Diarrhea (Gastrointestinal disorders) | 1 (6)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (6)
Inguinal hernia (Gastrointestinal disorders) | 1 (6)
Rectal polyp (Gastrointestinal disorders) | 1 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (6)
Adverse drug reaction (General disorders) | 1 (5)
Chest pain (General disorders) | 1 (5)
Death (General disorders) | 1 (5)
General physical health deterioration (General disorders) | 1 (5)
Unevaluable event (General disorders) | 1 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (13)
Cellulitis (Infections and infestations) | 1 (13)
Diverticulitis (Infections and infestations) | 1 (13)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (13)
Kidney infection (Infections and infestations) | 1 (13)
Labyrinthitis (Infections and infestations) | 1 (13)
Medical device site joint infection (Infections and infestations) | 1 (13)
Pneumonia (Infections and infestations) | 5 (13)
Sepsis (Infections and infestations) | 1 (13)
Urinary tract infection (Infections and infestations) | 2 (13)
Urosepsis (Infections and infestations) | 1 (13)
Wound infection (Infections and infestations) | 1 (13)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (10)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (10)
Fall (Injury, poisoning and procedural complications) | 3 (10)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (10)
Muscle strain (Injury, poisoning and procedural complications) | 1 (10)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (10)
Radius fracture (Injury, poisoning and procedural complications) | 1 (10)
Rib fracture (Injury, poisoning and procedural complications) | 1 (10)
Skin injury (Injury, poisoning and procedural complications) | 1 (10)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (10)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 1 (10)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (57)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (57)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (57)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (57)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (57)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (57)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (57)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (57)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 (57)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (57)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (57)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 (57)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (57)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (57)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (57)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (57)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (57)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (57)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (11)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (11)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (11)
Carpal tunnel syndrome (Nervous system disorders) | 1 (3)
Haemorrhagic stroke (Nervous system disorders) | 1 (3)
Occipital neuralgia (Nervous system disorders) | 1 (3)
Presyncope (Nervous system disorders) | 1 (3)
Confusional state (Psychiatric disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Joint prosthesis user (Social circumstances) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (4)
Hypotension (Vascular disorders) | 1 (4)
Peripheral artery occlusion (Vascular disorders) | 1 (4)
Varicose vein (Vascular disorders) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLOBAL ICON Stemless Shoulder System (N=156)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 2 (11)
Atrial fibrillation (Cardiac disorders) | 1 (11)
Bradycardia (Cardiac disorders) | 1 (11)
Cardiac failure (Cardiac disorders) | 1 (11)
Dilatation atrial (Cardiac disorders) | 1 (11)
Extrasystoles (Cardiac disorders) | 1 (11)
Heart valve incompetence (Cardiac disorders) | 1 (11)
Palpitations (Cardiac disorders) | 3 (11)
Silent myocardial infarction (Cardiac disorders) | 1 (11)
Tachycardia (Cardiac disorders) | 1 (11)
Ventricular extrasystoles (Cardiac disorders) | 1 (11)
Peutz-Jeghers syndrome (Congenital, familial and genetic disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Basedow's disease (Endocrine disorders) | 1 (2)
Goitre (Endocrine disorders) | 1 (2)
Age-related macular degeneration (Eye disorders) | 1 (11)
Cataract (Eye disorders) | 5 (11)
Diplopia (Eye disorders) | 1 (11)
Dry eye (Eye disorders) | 1 (11)
Entropion (Eye disorders) | 1 (11)
Epiretinal membrane (Eye disorders) | 1 (11)
Eye irritation (Eye disorders) | 1 (11)
Eye pain (Eye disorders) | 1 (11)
Macular degeneration (Eye disorders) | 1 (11)
Meibomian gland dysfunction (Eye disorders) | 1 (11)
Retinal haemorrhage (Eye disorders) | 1 (11)
Retinal tear (Eye disorders) | 1 (11)
Vitreous detachment (Eye disorders) | 1 (11)
Abdominal pain (Gastrointestinal disorders) | 1 (14)
Abdominal pain upper (Gastrointestinal disorders) | 1 (14)
Anal incontinence (Gastrointestinal disorders) | 1 (14)
Constipation (Gastrointestinal disorders) | 2 (14)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (14)
Dry mouth (Gastrointestinal disorders) | 1 (14)
Dysphagia (Gastrointestinal disorders) | 1 (14)
Gastritis (Gastrointestinal disorders) | 2 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (14)
Haematemesis (Gastrointestinal disorders) | 1 (14)
Hiatus hernia (Gastrointestinal disorders) | 1 (14)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (14)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (14)
Large intestine polyp (Gastrointestinal disorders) | 1 (14)
Nausea (Gastrointestinal disorders) | 2 (14)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (14)
Adverse drug reaction (General disorders) | 1 (18)
Catheter site inflammation (General disorders) | 1 (18)
Chest pain (General disorders) | 5 (18)
Early satiety (General disorders) | 1 (18)
Fatigue (General disorders) | 1 (18)
Gait disturbance (General disorders) | 1 (18)
Impaired healing (General disorders) | 2 (18)
Non-cardiac chest pain (General disorders) | 1 (18)
Pain (General disorders) | 2 (18)
Peripheral swelling (General disorders) | 3 (18)
Pyrexia (General disorders) | 2 (18)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (16)
Cellulitis (Infections and infestations) | 1 (16)
Cystitis (Infections and infestations) | 1 (16)
Diverticulitis (Infections and infestations) | 2 (16)
Erysipelas (Infections and infestations) | 1 (16)
Influenza (Infections and infestations) | 2 (16)
Lower respiratory tract infection (Infections and infestations) | 3 (16)
Onychomycosis (Infections and infestations) | 1 (16)
Pneumonia (Infections and infestations) | 1 (16)
Post procedural infection (Infections and infestations) | 2 (16)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (16)
Respiratory syncytial virus infection (Infections and infestations) | 1 (16)
Urinary tract infection (Infections and infestations) | 1 (16)
Viral infection (Infections and infestations) | 1 (16)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (24)
Back injury (Injury, poisoning and procedural complications) | 1 (24)
Bone contusion (Injury, poisoning and procedural complications) | 1 (24)
Burns second degree (Injury, poisoning and procedural complications) | 1 (24)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (24)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (24)
Chest injury (Injury, poisoning and procedural complications) | 1 (24)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (24)
Contusion (Injury, poisoning and procedural complications) | 1 (24)
Fall (Injury, poisoning and procedural complications) | 3 (24)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (24)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (24)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (24)
Joint injury (Injury, poisoning and procedural complications) | 1 (24)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (24)
Muscle strain (Injury, poisoning and procedural complications) | 1 (24)
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 1 (24)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (24)
Overdose (Injury, poisoning and procedural complications) | 1 (24)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (24)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (24)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (24)
Rib fracture (Injury, poisoning and procedural complications) | 1 (24)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (24)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (24)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (24)
Sternal Fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 (24)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (24)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (24)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (24)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (24)
Wound (Injury, poisoning and procedural complications) | 1 (24)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (24)
Crystal urine present (Investigations) | 1 (4)
HLA marker study positive (Investigations) | 1 (4)
Staphylococcus test positive (Investigations) | 1 (4)
Weight decreased (Investigations) | 1 (4)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (4)
Gout (Metabolism and nutrition disorders) | 1 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (69)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (69)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (69)
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 (69)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (69)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (69)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (69)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (69)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (69)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (69)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (69)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (69)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (69)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (69)
Joint noise (Musculoskeletal and connective tissue disorders) | 2 (69)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 (69)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (69)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (69)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (69)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (69)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (69)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (69)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (69)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (69)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (69)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 25 (69)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (69)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (69)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (69)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 (69)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (69)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (69)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (69)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (69)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (69)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (12)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (12)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (12)
Acquired syringomyelia (Nervous system disorders) | 1 (24)
Carpal tunnel syndrome (Nervous system disorders) | 7 (24)
Dizziness (Nervous system disorders) | 2 (24)
Headache (Nervous system disorders) | 1 (24)
Hypoaesthesia (Nervous system disorders) | 3 (24)
Lumbar radiculopathy (Nervous system disorders) | 1 (24)
Memory impairment (Nervous system disorders) | 1 (24)
Migraine (Nervous system disorders) | 1 (24)
Neuralgia (Nervous system disorders) | 1 (24)
Neuropathy peripheral (Nervous system disorders) | 1 (24)
Paraesthesia (Nervous system disorders) | 3 (24)
Pseudoradicular syndrome (Nervous system disorders) | 1 (24)
Sensory loss (Nervous system disorders) | 1 (24)
Spinal claudication (Nervous system disorders) | 2 (24)
Transient ischaemic attack (Nervous system disorders) | 1 (24)
Device loosening (Product Issues) | 1 (1)
Delirium (Psychiatric disorders) | 1 (3)
Depression (Psychiatric disorders) | 1 (3)
Panic attack (Psychiatric disorders) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (6)
Haematuria (Renal and urinary disorders) | 1 (6)
Hydronephrosis (Renal and urinary disorders) | 1 (6)
Pollakiuria (Renal and urinary disorders) | 1 (6)
Urinary incontinence (Renal and urinary disorders) | 1 (6)
Urinary retention (Renal and urinary disorders) | 1 (6)
Urinary tract pain (Renal and urinary disorders) | 1 (6)
Breast disorder (Reproductive system and breast disorders) | 1 (4)
Breast pain (Reproductive system and breast disorders) | 1 (4)
Breast swelling (Reproductive system and breast disorders) | 1 (4)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (12)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (11)
Blister (Skin and subcutaneous tissue disorders) | 1 (11)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (11)
Rash (Skin and subcutaneous tissue disorders) | 1 (11)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (11)
Skin lesion (Skin and subcutaneous tissue disorders) | 4 (11)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (11)
Aortic aneurysm (Vascular disorders) | 1 (9)
Haematoma (Vascular disorders) | 6 (9)
Hypertension (Vascular disorders) | 1 (9)
Peripheral coldness (Vascular disorders) | 1 (9)

LIMITATIONS AND CAVEATS:
Due to investigators decision study was terminated at 5 years. Therefore, results are reported only up to 5 years (60 months).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03168672/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT03168672/SAP_001.pdf